CLINICAL TRIAL: NCT01629537
Title: A Randomized, Placebo-Controlled Trial of Stellate Ganglion Block in the Treatment of Post Traumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven Hanling, Department of Psychaitry Research Director, Mental Health Directorate, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NMCSD.2010.0157
Record Dates: First submitted 2012-06-22; First posted 2012-06-27 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Post Traumatic Stress Disorder (PTSD)
Keywords: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Other): Subjects 1 month post in the placebo group who demonstrate either the same level of PTSD severity at enrollment or worsening of the condition (i.e., CAPS score greater than or equal to 40) will be offered SGB treatment and crossed over to active treatment. Patients who cross over from placebo to active SGB treatment will be followed one week, one month and three months after cross over.
  Interventions: Procedure: Placebo Procedure
- Stellate Ganglion Block (SGB) (Experimental): Subjects assigned to SGB arm will undergo SGB procedure and be followed one week, one month and three months after procedure or until CAPS score is below 40.
  Interventions: Procedure: Stellate Ganglion Block injection with ropivicane

INTERVENTIONS:
Procedure: Stellate Ganglion Block injection with ropivicane — For participants receiving the stellate ganglion injection with ropivicaine, a 22 g needle will be directed percutaneously to the anterolateral C6 vertebral body Using ultrasound guidance to avoid the nearby vascular structures and identify the appropriate vertebral level and tissue plane. After negative aspiration for blood and CSF, and digital subtraction, 2cc of Iohexol,(Omnipaque 180) will be injected through the needle under live fluoroscopy to visualize dye spread over the pre-vertebral plane At this point, 7 cc 0.5% ropivicaine will be injected and the needle will be removed.
  Arms: Stellate Ganglion Block (SGB)
Procedure: Placebo Procedure — In participants randomized to the placebo injection, the same positioning, monitoring, sterile preparation and technique and local anesthesia protocol will be used. The 22 g needle will instead be placed in the subcutaneous, superficial tissues overlying the C6 tubercle, but superficial enough that the prevertebral fascial plane of the stellate ganglion will not be breached. Using fluoroscopic guidance, this needle will be injected with 2 cc of contrast dye to confirm superficial spread. The needle will then be injected with 5 cc of preservative free normal saline and the needle will be removed.
  Arms: Placebo

SUMMARY:
Post Traumatic Stress Disorder (PTSD), is a devastating condition which causes distress or impairment in social, occupational or other important aspects of functioning. The occurrence of PTSD in the military is on the rise. This has significantly impacted military members, their families, and society as a whole. According to an expert panel convened by the Institute of Medicine in 2007, the effectiveness of most currently employed PTSD therapies is low. Safe and effective treatments are urgently needed. The specific aim of this investigation is to evaluate the effectiveness of a novel approach to relieve PTSD symptoms, utilizing a procedure commonly used in pain management, a Stellate Ganglion Block (SGB) with local anesthesia. Male soldiers experiencing moderate to severe symptoms of PTSD will be recruited for evaluation of Stellate Ganglion Block with local anesthesia as an intervention for PTSD treatment. Participants will be randomized to receive either the SGB with local anesthesia to C6 tubercle or a sham procedure involving a subcutaneous saline injection to the neck. The PTSD symptoms before and after the procedure will be measured using a comprehensive clinician-administered scale, self-report measures, objective measures of cognitive ability, and physiologic reactivity measures. Subjects will undergo assessment prior to the procedure, one week following the procedure, one month and 3 months following the procedure. Patients receiving sham injections will be allowed to cross over to the treatment group. Based on published case reports of Lipov et al in Chicago and Mulvaney et al from Walter Reed Medical Center, who utilized this technique to successfully treat soldiers with combat-related PTSD, we predict that the use of Stellate Ganglion Block will result in reduction of PTSD symptoms as measured by clinician-administered scales, self-report measures, objective measures of cognitive ability, and physiologic reactivity measures, leading to a significant and lasting reduction of PTSD symptoms.

ELIGIBILITY:
1. Gender: Male and Female
2. Minimum Age/ Maximum Age: Over the age of 18
3. Accepts Healthy Volunteers:

Yes, but must be experiencing mild to severe symptoms of PTSD

Inclusion Criteria will include subjects who:

* Subjects, (male and/or female), experiencing moderate-to-severe PTSD Symptoms
* Subjects, (male and/or female), who elect to undergo the SGB procedure.
* DEERS Eligible

Exclusion Criteria will include subjects who:

* Have an acute, unstable medical condition i.e., temperature, blood pressure, heart rate outside normal limits; electrolyte abnormalities; mental conditions which preclude informed consent/unable to make decisions independently; on antibiotic therapy; uncontrolled seizures; nausea/vomiting; night sweats; blood dyscrasias.
* Have acute infections or cardiac compromise or irregularities of heart rate or rhythm.
* Pathologic bradycardia
* Have local infections of the anterior neck region
* Have severe pulmonary disease, (in severe pulmonary disease, the patient may experience severe shortness of breath on minimal exertion [even at rest], require supplemental oxygen, is progressively disabled and may have a constant cough and associated wheeze).
* Are anticoagulated
* Have a blood clotting disorder
* Have an American Society of Anesthesiologists (ASA) physical status score of 3 or higher (severe systemic disease, not incapacitating)
* Have allergic reactions to local anesthetics and / or contrast dyes,
* Have conditions or disorders that affect cognitive functioning, including stroke, past or present diagnosis of psychosis,
* Have conditions that invalidate testing procedures (e.g., English not first language, inability to write, speak, read, etc.)
* Have Horner's syndrome on the right side
* Have a diagnosis of glaucoma
* Are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2011-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PSTD Scale (CAPS) | 1 week
  The CAPS is generally considered the gold standard for PTSD assessment, and will be used to determine severity of PTSD symptoms compared to the 1 week pre baseline measures at enrollment

SECONDARY OUTCOMES:
PTSD Checklist Military Version (PCL-M) | 1 week
  The PCL is a 17-item self-report measure of the 17 DSM-IV symptoms of PTSD. It is used to screen and diagnose individuals for PTSD, as well as monitoring symptom change during and after treatment. To be compared to the 1 week pre baseline measures at enrollment
The Patient Health Questionnaire 9 (PHQ-9) | 1 week
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. To be compared to the 1 week pre baseline measures at enrollment
Beck Anxiety Inventory (BAI) | 1 week
  A 21-question multiple-choice self-report inventory that is used for measuring the severity of an individual's anxiety. To be compared to the 1 week pre baseline measures at enrollment
Sheehan Disability Scale (SDS) | 1 week
  Assesses disability in work/school activities, family relationships, and social functioning, and it evaluates the functional impact of psychiatric disorders. To be compared to the 1 week pre baseline measures at enrollment
Behavioral Reactivity Test (BRT) | 1 week
  To be compared to the 1 week pre baseline measures at enrollment
Automated Neuropsychological Assessment Metric (ANAM) | 1 week
  Computer-based assessments of cognitive domains including attention, concentration, reaction time, memory, processing speed, and decision-making. Evaluate changes in an individual's cognitive status over time. To be compared to the 1 week pre baseline measures at enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hanling, MD, CDR, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- United States Naval Medical Center San Diego, San Diego, California, United States